CLINICAL TRIAL: NCT06261216
Title: Association Between Lifetime Physical Activity and Exercise and the Development of Wild-type Transthyretin Amyloid Cardiomyopathy
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 01/2023/LPA-wtATTR/NVNS
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Amyloid Cardiomyopathy; Wild Type ATTR Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 40mL of blood in aliquots at -80°C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- wild-type transthyretin amyloid cardiomyopathy
  Interventions: Other: Interview
- heart failure
  Interventions: Other: Interview
- healthy controls
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — * International Physical Activity Questionnaire (IPAQ-SF)
  * interviewer-administered modified Lifetime Total Physical Activity Questionnaire (LTPAQ) form

SUMMARY:
The aim of this study is to investigate the association between increased lifetime physical activity and the development of wild-type transthyretin amyloid cardiomyopathy.

DETAILED DESCRIPTION:
Transthyretin amyloidosis is considered to be the most common cause of cardiac amyloidosis, with an increasing diagnosis rate over the last decade. Though once considered to be a rare disease, recent data suggest it is underappreciated as a common cause of cardiac diseases and syndromes such as left ventricular hypertrophy, aortic stenosis, and heart failure with preserved ejection fraction, especially in the elderly. Wild-type transthyretin amyloidosis, which is associated with ageing, is currently considered to be the most frequent form of amyloidosis worldwide, and is dominated by cardiac symptoms. Other than male gender and advanced age, risk factors for the development of wild-type transthyretin amyloid cardiomyopathy (wtATTR-CM) are largely unknown. There is rising empirical observation that patients with wtATTR-CM frequently have a substantial history of athletic activity, which might contribute to the manifestation of the disease.

This study aims to create evidence of a correlation between increased lifetime physical activity and the development of wtATTR-CM. Furthermore, the investigators aim to explore the association between certain sport disciplines and disease development.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of wtATTR-CM including sequencing of the TTR gene; or HF; or healthy proband without a diagnosis of heart disease
2. Initial diagnosis of respective cardiac disease (wtATTR-CM, HF) after the 6th decade of life; or no cardiac disease (healthy control)
3. Willingness and ability to provide signed informed consent form (ICF)
4. Age > 60 years

Exclusion Criteria:

1. History of severe chronic illness limiting the ability to perform physical activity during the 3rd to 6th decade
2. A diagnosis of dementia or cognitive impairment
3. Any other reason resulting in the inability to perform the questionnaire and/or interview
4. Known disease-causing variant (pathogenic or likely-pathogenic) in the TTR gene

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Number of participants: 189 The study population will comprise three subgroups (n=63 in each group)
  1. cardiac wild type transthyretin amyloidosis (wtATTR-CM);
  2. heart failure (HF);
  3. healthy individuals without heart disease
Sampling Method: Non-Probability Sample
Enrollment: 189 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Association between lifetime physical activity (in METs) and disease development | 3rd to 6th decade
  Association between lifetime physical activity (in METs per active decade) and the development of wild-type transthyretin amyloid cardiomyopathy

SECONDARY OUTCOMES:
Association between lifetime athletic activity (in METs) and disease development | 3rd to 6th decade
  Association between lifetime athletic activity (in METs per active decade) and the development of wild-type transthyretin amyloid cardiomyopathy

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Verheyen, Res Prof, MD PhD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No